CLINICAL TRIAL: NCT03748693
Title: Inflammation and Cellular Immunity in Vaginal Tissue in Patients With Pelvic Organ Prolapse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0073-18
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POP Group: Women with POP undergoing surgery in our OB/GYN department.
  Interventions: Procedure: Colporrhaphy
- Non-POP Group: Women undergoing hysterectomy for other indications.
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Surgery performed on women with a variety of gynecological indications
  Groups: Non-POP Group
Procedure: Colporrhaphy — Surgery performed on women with POP
  Groups: POP Group

SUMMARY:
The aim of this study is to investigate the inflammatory and maturation processes of immature myeloid cells (IMC) in the vaginal tissue in women with advanced pelvic organ prolapse (POP) (stage III-IV) and in normal non-POP controls.

We hypothesize that the processes contributing to POP may be related to immune response and changes in myeloid cell populations and the cytokine environment.

ELIGIBILITY:
Inclusion Criteria:

* Women with POP undergoing colporrhaphy
* Women undergoing hysterectomy

Exclusion Criteria:

* Autoimmune and connective tissue disorders
* Cancer in genital tract

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women attending our OB/GYN department because of POP and other gynecological disorders
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Immune response in POP | Two weeks
  Tissue biopsy will analyzed for IMC and compared to control group
Cytokine environment in POP | Two weeks
  Tissue biopsy will analyzed for cytokine environment and compared to control group

IPD SHARING:
Plan to Share IPD: No